CLINICAL TRIAL: NCT03823248
Title: Therapeutic Mechanism of Jianpi Huoxue Recipe in Treating Gastric Premalignant Lesion：A Multi-center, Randomized and Controlled Experiment
Brief Title: Jianpi Huoxue Recipe in Treating Gastric Premalignant Lesion
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xiyuan Hospital of China Academy of Chinese Medical Sciences (Other)
Collaborators: Guangdong Provincial Hospital of Traditional Chinese Medicine (Other); Beijing Friendship Hospital (Other); Wuhan Integrated Traditional Chinese and Western Medicine Hospital (Other); The Second Affiliated Hospital of Tianjin University of Traditional Chinese Medicine (Unknown); The Second Affiliated Hospital of Hunan University of Traditional Chinese Medicine (Other); The Affiliated Hospital of Shaanxi University of Traditional Chinese Medicine (Unknown); Traditional Chinese Medicine Hospital of KUNSHAN (Unknown); Yueyang Hospital of Integrated Traditional Chinese and Western Medicine (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2017YFC1700601
Record Dates: First submitted 2018-07-11; First posted 2019-01-30 (Actual); Last update posted 2021-06-25 (Actual); Status verified 2021-06

CONDITIONS: Gastric Precancerous Condition
MeSH Terms: interventions — moluodan; Folic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MoLuoDan and Sanchi powder group (Experimental): Experiment group: oral administration of Moluodan concentrated pills with warm water before meal for 8 pills each time for three times a day, + oral administration of Sanchi powder mixing with warm water before meal for 3g each time for twice a day, + oral administration of Folic Acid Tablet simulation half a hour after meal for 5 mg each time for 3 times a day. The medication period was 24 weeks.
  Interventions: Drug: MoLuoDan; Drug: Sanchi powder; Drug: Folic Acid Tablet simulation
- Folic Acid Tablet group (Active Comparator): Control group: oral administration of Moluodan simulation medicine with warm water before meal for 8 pills each time for three times a day, + oral administration of Sanchi powder simulation medicine mixing with warm water before meal for 3g each time for twice a day, + oral administration of folic acid tablets half a hour after meal for 5 mg each time for 3 times a day. The medication period was 24 weeks.
  Interventions: Drug: Folic Acid Tablet; Drug: MoLuoDan simulation; Drug: Sanchi powder simulation

INTERVENTIONS:
Drug: MoLuoDan — oral administration of Moluodan concentrated pills with warm water before meal for 8 pills each time for three times a day
  Arms: MoLuoDan and Sanchi powder group
Drug: Sanchi powder — oral administration of Sanchi powder mixing with warm water before meal for 3g each time for twice a day
  Arms: MoLuoDan and Sanchi powder group
Drug: Folic Acid Tablet — oral administration of folic acid tablets half an hour after meal for 5 mg each time for 3 times a day.
  Arms: Folic Acid Tablet group
Drug: MoLuoDan simulation — oral administration of Moluodan simulation medicine with warm water before meal for 8 pills each time for three times a day
  Arms: Folic Acid Tablet group
Drug: Sanchi powder simulation — oral administration of Sanchi powder simulation medicine mixing with warm water before meal for 3g each time for twice a day
  Arms: Folic Acid Tablet group
Drug: Folic Acid Tablet simulation — oral administration of folic acid simulation tablets half a hour after meal for 5 mg each time for 3 times a day.
  Arms: MoLuoDan and Sanchi powder group

SUMMARY:
This study had adopted the multi-center, randomized and controlled experiment design based on standardized mucosal biopsy and pathohistological operation, as well as therapeutic evaluation methodology. Meanwhile, patients diagnosed with chronic atrophic gastritis accompanying with low grade intraepithelial neoplasia and indefinite dysphasia (grade C2/C3 of Vienna classification) confirmed by gastroscopic histopathology were enrolled as the objects of study, while folic acid was used as the control. The therapeutic effect and safety of Jianpi Huoxue Recipe (Moluodan + Sanchi powder) in intervening the gastric Premalignant lesion were evaluated from the points of view of pathology, gastroscopy and symptoms. The elimination rate of intraepithelial neoplasia of gastric mucosa was expected to be improved by 9-12%. Moreover, high quality evidence-based medical evidence regarding traditional Chinese medicine (TCM) in intervening gastric Premalignant lesion would be obtained, which could form the mature, propagable and effective scheme.

DETAILED DESCRIPTION:
Intraepithelial neoplasia of gastric mucosa is a well-recognized gastric Premalignant lesion, which is the key of secondary prevention for gastric cancer. However, no universally acknowledged effective therapeutic scheme is available at present. Previously, the investigator's research group has carried out clinical trial study based on solving the key problems such as diagnostic criteria, mucosal biopsy consistency and therapeutic evaluation methodology, and has attained certain achievements. This study had adopted the multi-center, randomized and controlled experiment design based on standardized mucosal biopsy and pathohistological operation, as well as therapeutic evaluation methodology. Meanwhile, patients diagnosed with chronic atrophic gastritis accompanying with low grade intraepithelial neoplasia and indefinite dysphasia (grade C2/C3 of Vienna classification) confirmed by gastroscopic histopathology were enrolled as the objects of study, while folic acid was used as the control. The therapeutic effect and safety of Jianpi Huoxue Recipe (Moluodan + Sanchi powder) in intervening the gastric Premalignant lesion were evaluated from the points of view of pathology, gastroscopy and symptoms. The elimination rate of intraepithelial neoplasia of gastric mucosa was expected to be improved by 9-12%. Moreover, high quality evidence-based medical evidence regarding traditional Chinese medicine (TCM) in intervening gastric Premalignant lesion would be obtained, which could form the mature, propagable and effective scheme. At the same time, molecular and biological indicators, including CDX2, SOX2, MUC2, MUC6, MUC5AC and CD10, were detected using the pathological tissues, so as to explore the therapeutic mechanism of Jianpi Huoxue Recipe in intervening gastric Premalignant lesion, and to construct the model platform for special disease research on gastric Premalignant lesion.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatients and inpatients diagnosed with chronic atrophic gastritis accompanying with low grade intraepithelial neoplasia and indefinite dysphasia confirmed by gastroscopy and histopathological examination;
2. Patients aged from 18-75 years;
3. Subjects who were informed and voluntarily signed the informed consent.

Exclusion Criteria:

1. Patients pathohistologically diagnosed with high grade intraepithelial neoplasia/severe dysplasia;
2. Patients with a history of gastric ulcer, gastric polyps and gastric surgery;
3. Patients taking NSAIDs for a long term;
4. Patients suspected of gastric cancer or malignant lesions in other systems;
5. Patients with a history of gastric surgery;
6. Patients with concurrent primary diseases in cardiovascular, cerebrovascular, liver, kidney and hemopoietic systems (ALT>80 u/L, and/or AST>80 u/L, with abnormal renal function)
7. Patients with mental disease, dysgnosia and logopathy;
8. Pregnant women, or those preparing a pregnancy and breastfeeding women;
9. Patients with a allergic history of medicines used in this experiment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
The disappearance rate of dysplasia | six months
  The all patients' histopathology will be evaluated two times, the first time is when the patients' are included into the clinical trials, the second time is after 24 weeks treatment in each group, patients' histopathology should be evaluated for comparison between two groups,at the same time patients' histopathology should be evaluated for comparison in each group.The change in histological score (mean score of all biopsie after treatment in each group and between groups was calculated. The response rate of each pathological lesion was calculated as a percentage of those improved or disappeared at the 6th month to all subjects. The disappearance rate of dysplasia between groups were compared, which was defined as the absence of dysplasia (score 0) in all biopsy specimens after treatment.
The score changes of histopathology | six months
  The score changes of atrophy, intestinal metaplasia, chronic inflammation and active inflammation compared between baseline and after 6-month treatment.

SECONDARY OUTCOMES:
The score changes of Endoscopic Findings | six months
  The score changes of endoscopic findings, such as erosion, bleeding, coarse and uneven mucosa, and bile reflux were compared between baseline and after 6-month treatment.
Main symptom score | six months
  Changes of symptom score were compared. The symptom include upper abdominal pain, upper abdominal distension, poor appetite, nausea and belching. The disappearance rate of symptom was expressed as a percentage of the subjects whose symptoms disappeared after medication to those exhibiting symptoms before medication.
The patient-reported outcome (PRO)scale integrals | six months
  The patient-reported outcome (PRO) instrument for chronic gastrointestinal diseases was a 35-item instrument, including 6 dimensions of regurgitation, dyspepsia, defecation, general condition, emotion and social function. All items graded into 5 levels and scored 0-4, except for decreased appetite, which is grouped into 4 levels and scored 0-3.

CONTACTS AND LOCATIONS:
Locations (1):
- Xiyuan Hospital of China Academy of Chinese Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: No